CLINICAL TRIAL: NCT00892619
Title: Comparison of Two Techniques for Epiretinal or Internal Limiting Membrane Peel.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: PETROS EUTHYMIOU CARVOUNIS, M.D., Baylor College of Medicine, Micheal Debakey Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: h-22378
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-04

CONDITIONS: Epiretinal Membrane; Vitreomacular Traction
Keywords: Epiretinal Membrane; Vitreomacular traction; MVR blade; Tano brush; ILM forceps; surgical technique
MeSH Terms: conditions — Epiretinal Membrane | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILM forceps (Experimental): Using ILM forceps to initiate and complete peel
  Interventions: Procedure: using ILM forceps alone
- Other (Active Comparator): Using an instrument to create a break in the ILM followed by peeling of the membrane with end-grasping forceps
  Interventions: Procedure: Breaking and peeling with end-grasping forceps

INTERVENTIONS:
Procedure: using ILM forceps alone — Using ILM forceps to initiate and complete ILM peel
  Arms: ILM forceps
Procedure: Breaking and peeling with end-grasping forceps — Using an instrument to create a break in the ILM followed by peeling of the membrane with end-grasping forceps
  Arms: Other

SUMMARY:
Epiretinal membranes (ERM) are cellular membranes on the surface of the retina that result in distortion of the vision (metamorphopsia), and decreased best-corrected visual acuity. They are most frequently found in patients over the age of 50 and have a reported prevalence of 7-12%. [1,2] Epiretinal membranes are caused by posterior vitreous separation, retinal detachment, proliferative vitreoretinopathy, cataract surgery, trauma, inflammation, retinal vascular disease, and idiopathic. [1-4] Epiretinal membrane removal by pars plana vitrectomy combined with internal limiting membrane peeling leads to improved vision, decreased metamorphopsia, and improved quality of life after surgery. [2] Internal limiting membrane (ILM) peel has been associated with decreased rates of epiretinal membrane recurrence and is also performed during vitrectomy for repair of macular holes or vitreomacular traction. [5,6] Internal limiting membrane peeling can be performed by using an instrument to make a break in the membrane followed by peeling with forceps, or by utilizing ILM forceps alone to pinch and peel an unviolated ILM. No study exists comparing different intraoperative techniques used for ILM peeling on visual outcomes and operating time. The investigators hypothesize that using a "pinch and peel" technique will equal outcomes with shorter operating time than other techniques.

1. McDonald HR, Johnson RN, Ai E, Jumper JM, Fu AD. Macular epiretinal membranes. Retina, 4th edition, editor Ryan SJ, Wilkinson CP, 2006, p 2509-2525.
2. Ghazi-Nouri SM, Tranos PG, Rubin GS, Adams ZC, Charteris DG. Vitrectomy and epiretinal membrane peel surgery visual function and quality of life following. 2006;90;559-562; Br. J. Ophthalmol
3. Haritoglu C, Gandorfer A, Gass CA, Schaumberger M, Ulbig MW, Kampik A. The Effect of Indocyanine-Green on Functional Outcome of Macular Pucker Surgery. AM. J. Ophthal. VOL. 135,NO.3, 328-337, Mar 2003
4. Hiscott PS, Grierson I, McLeod D. Retinal pigment epithelial cells in epiretinal membranes: an immunohistochemical study. Br. J. Ophthalmol, 1984, 68, 708-715
5. Park DW, Dugel PU, Garda J, Sipperley JO, Thach A, Sneed SR, Blaisdell J. Macular Pucker Removal with and without Internal Limiting Membrane Peeling: Pilot Study. Ophthalmology Volume 110, 1, Jan 2003
6. Kwok AK, Lai TY, Yuen KS. Epiretinal membrane surgery with or without internal limiting membrane peeling. Clinical and Experimental Ophthalmology, 2005, 33:379-385

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal membrane with associated macular thickening or cystoid macular edema present;
* ETDRS best corrected visual acuity 20/50 or worse attributed to the effects of the epiretinal membrane;
* Pars plana vitrectomy/membrane peel planned for treatment of the epiretinal membrane;
* Patients older than 19 years of age;
* No co-existent retina pathology or optic neuropathy that may influence the visual field.

Exclusion Criteria:

* Patient unwilling or unable to provide informed consent;
* Co-existing retina pathology (proliferative diabetic retinopathy, central retinal vein occlusion, branch retinal vein occlusion, central/branch retinal artery occlusion, ERM secondary to trauma, prior surgery for ERM);
* Co-existing lenticular opacity;
* Optic neuropathy causing a pre-existing visual field defect involving the central 10 degrees of vision.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2008-12; Primary Completion 2010-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity | three months

SECONDARY OUTCOMES:
Change in humphrey visual field | three months

CONTACTS AND LOCATIONS:
Overall Officials: Petros E Carvounis, B.M.B.Ch., F.R.C.S.C., Principal Investigator — Baylor College of Medicine, Michael Debakey VAMC
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Michael Debakey VAMC, Houston, Texas